CLINICAL TRIAL: NCT02807142
Title: Efficacy Assessment of the Cell Therapy Medicine NC1 in Patients With Post-traumatic Syringomyelia
Acronym: CME-LEM4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Jesús Vaquero Crespo, M.D., M.D., Puerta de Hierro University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CME-LEM4
Record Dates: First submitted 2016-06-03; First posted 2016-06-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Post-Traumatic Syringomyelia
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NC 1 cell therapy (Experimental): All patients will be treated with the same treatment: NC1 cell therapy
  Interventions: Biological: NC 1 cell therapy

INTERVENTIONS:
Biological: NC 1 cell therapy — All patients will be treated with NC1

SUMMARY:
The objective of the study is to determine if the cell therapy NC1 administered in the spinal cord is effective for the treatment of a post-traumatic syringomyelia. The post-traumatic syringomyelia is the development and progression of cyst filled with cerebrospinal fluid (CSF) within the spinal cord. The cell therapy NC1 consist on cells obtained from the bone marrow of the patient, that are cultured in vitro and administered in the spinal cord of the same patient.

DETAILED DESCRIPTION:
Phase II, Open, prospective, not controlled, not randomized clinical trial in patients affected by post-traumatic syringomyelia. The trial evaluates the efficacy of the cell therapy NC1 administered via intrathecal in the location of the injury. After the administration of the cell therapy, patients will undergo physiotherapy during the follow-up period (6 months). Patients will be evaluated at month 3 and month 6 after the NC1 administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with traumatic medullar injury (levels A, B, C or D of the ASIA scale) and associated syringomyelia in at least three spinal segments, and with neurological deficit clinically stable at least 6 months prior to treatment.
* Previous studies in Neurophysiology, MR, Urology (if data on neurogenic bowel exists), defecatory function (if data on neurogenic intestine exists)
* Age between 18 and 70 years old.
* Presence of syringomyelia based on a neuro-image (MR)
* Patients will compromise to use anticonceptive measures from the cell extraction until 6 months after the administration of the treatment.
* Patients will compromise to a clinical follow-up and to perform physical therapy, one hour daily five days per week during the treatment period.
* Patients should sign an written informed consent.
* Haematological and creatinin parameters, SGOT and SGPT into the normal ranges.

Exclusion Criteria:

* Patients under 18 or above 70 years old
* Pregnancy or breastfeeding
* Neoplasia in the last 5 years
* Patients with systemic diseases that increase the risk of the surgical intervention
* Genetics alterations that could conduct to cellular transformation during the cellular expansion phase.
* Patients not really sure of their cooperation to follow the physical therapy or clinical controls during the study.
* Additional neurodegenerative diseases
* Drug consuming, psychiatric disease or allergy to proteins used during cellular expansion
* HIV or syphilis positive serologies
* Active Hepatitis B or c, based on serologies
* Any other reasons according to the investigator criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03; Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of the treatment with NC1 in terms of improvement of neurological sequelae in patients with post traumatic syringomyelia using the ASIA scale (American Spinal Injury Association | Pretreatment, month 3 post treatment, month 6 post treatment
  Neurological evaluation is done using ASIA scale (American Spinal Injury Association)

SECONDARY OUTCOMES:
Safety, by the assessment of the adverse events of the study | 1 year
  Adverse events
Efficacy of the treatment with NC1 in terms of improvement of neurological sequelae in patients with post traumatic syringomyelia assessed with the IANR-SCIFRS scale (Injury Functional Rating Scale) | Pretreatment, month 3 post treatment, month 6 post treatment
  Neurological evaluation is done using IANR-SCIFRS scale (Injury Functional Rating Scale)
Efficacy of the treatment with NC1 in terms of improvement of neurological sequelae in patients with post traumatic syringomyelia in terms of spams frequency | Pretreatment, month 3 post treatment, month 6 post treatment
  Neurological evaluation is done using PENN scale (spams frequency score)
Efficacy of the treatment with NC1 in terms of improvement of neurological sequelae in patients with post traumatic syringomyelia in term of spasticity | Pretreatment, month 3 post treatment, month 6 post treatment
  Neurological evaluation is done using Ashworth scale (spasticity)
Efficacy of the treatment with NC1 in terms of improvement of neurological sequelae in patients with post traumatic syringomyelia using the Visual Analog Scale | Pretreatment, month 3 post treatment, month 6 post treatment
  Neurological evaluation is done using EVA scale (Visual Analog Scale)
Efficacy of the treatment with NC1 in terms of improvement of neurological sequelae in patients with post traumatic syringomyelia in terms of bladder functionality | Pretreatment, month 3 post treatment, month 6 post treatment
  Neurological evaluation is done using GEFFNER scale (bladder functionality)
Efficacy of the treatment with NC1 in terms of improvement of neurological sequelae in patients with post traumatic syringomyelia using the Behavior Dimensions Scale | Pretreatment, month 3 post treatment, month 6 post treatment
  Neurological evaluation is done using BDS scales (Behavior Dimensions Scale)
Efficacy of the treatment with NC1 in terms of improvement of neurological sequelae in patients with post traumatic syringomyelia in terms of somatosensory or motor evoked potentials | Pretreatment, month 3 post treatment, month 6 post treatment
  Present of somatosensory or motor evoked potentials
Efficacy of the treatment with NC1 in terms of improvement of neurological sequelae in patients with post traumatic syringomyelia by electromyography | Pretreatment, month 3 post treatment, month 6 post treatment
  EMG (Electromyography)
Efficacy of the treatment with NC1 in terms of improvement of neurological sequelae in patients with post traumatic syringomyelia studying the spinal cord morphology | Pretreatment, month 3 post treatment, month 6 post treatment
  Spinal cord morphology (by Magnetic Resonance)
Efficacy of the treatment with NC1 in terms of improvement of neurological sequelae in patients with post traumatic syringomyelia in terms of defecatory function | Pretreatment, month 3 post treatment, month 6 post treatment
  Neurological evaluation is done assessing the defecatory function

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Vaquero Crespo, M.D., Principal Investigator — Hospital Universitario Puerta de Hierro-Majadahonda

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual data of participants will be shared with Authorities at the end of the Clinical Development Plan by the CTD (Common Technical Document). Results will be published in a scientific publication.
Time Frame: Starting at CTD submission to authorities.
Access Criteria: Spanish competent authority.

REFERENCES:
- [Background] Vaquero J, Zurita M. Bone marrow stromal cells for spinal cord repair: a challenge for contemporary neurobiology. Histol Histopathol. 2009 Jan;24(1):107-16. doi: 10.14670/HH-24.107. PMID 19012250
- [Background] Vaquero J, Zurita M. Functional recovery after severe CNS trauma: current perspectives for cell therapy with bone marrow stromal cells. Prog Neurobiol. 2011 Mar;93(3):341-9. doi: 10.1016/j.pneurobio.2010.12.002. Epub 2010 Dec 14. PMID 21163325
- [Background] Otero L, Zurita M, Bonilla C, Aguayo C, Rico MA, Rodriguez A, Vaquero J. Allogeneic bone marrow stromal cell transplantation after cerebral hemorrhage achieves cell transdifferentiation and modulates endogenous neurogenesis. Cytotherapy. 2012 Jan;14(1):34-44. doi: 10.3109/14653249.2011.608349. Epub 2011 Sep 23. PMID 21942842
- [Background] Otero L, Zurita M, Bonilla C, Aguayo C, Vela A, Rico MA, Vaquero J. Late transplantation of allogeneic bone marrow stromal cells improves neurologic deficits subsequent to intracerebral hemorrhage. Cytotherapy. 2011 May;13(5):562-71. doi: 10.3109/14653249.2010.544720. Epub 2011 Jan 5. PMID 21208021
- [Background] Huang H, Xi H, Chen L, Zhang F, Liu Y. Long-term outcome of olfactory ensheathing cell therapy for patients with complete chronic spinal cord injury. Cell Transplant. 2012;21 Suppl 1:S23-31. doi: 10.3727/096368912X633734. PMID 22507677